CLINICAL TRIAL: NCT03367013
Title: Lactoferrin Infant Feeding Trial - LIFT_Canada
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Elizabeth Asztalos (Other)
Collaborators: Sunnybrook Research Institute (Toronto, Ontario) (Unknown); Canadian Institutes of Health Research (CIHR) (Other Government); National Health and Medical Research Council, Australia (Other)
Responsible Party: Sponsor-Investigator, Dr. Elizabeth Asztalos, Neonatologist, Sunnybrook Health Sciences Centre
Organization: Sunnybrook Health Sciences Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 0890
Record Dates: First submitted 2017-12-04; First posted 2017-12-08 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Preterm Infant; Very Low Birth Weight Infant; Morbidity;Newborn
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): The intervention group will receive a daily dose of 200 mg/kg of bovine lactoferrin in breast/donor human milk or formula milk until 34 weeks corrected gestation or for a minimum of 2 weeks, whichever is longer, or until discharge home or transfer, if earlier.
  Interventions: Dietary Supplement: Bovine Lactoferrin
- Control Group (Sham Comparator): The control group will receive daily study feed with no bovine lactoferrin added in breast/donor human milk or formula milk until 34 weeks corrected gestation or for a minimum of 2 weeks, whichever is longer, or until discharge home or transfer, if earlier.
  Interventions: Other: No Bovine Lactoferrin added

INTERVENTIONS:
Dietary Supplement: Bovine Lactoferrin — Intervention includes a daily dose of 200 mg/kg bovine lactoferrin in breast/donor human milk or formula milk until 34 weeks corrected gestation or for a minimum of 2 weeks, whichever is longer, or until discharge home or transfer, if earlier.
  Other Names: Lactoferrin-250
  Arms: Intervention Group
Other: No Bovine Lactoferrin added — Control includes daily study feed with no bovine lactoferrin added in breast/donor human milk or formula milk until 34 weeks corrected gestation or for a minimum of 2 weeks, whichever is longer, or until discharge home or transfer, if earlier.
  Arms: Control Group

SUMMARY:
This is a multicentre, phase III, 2-arm, masked randomized controlled trial. The primary hypothesis is that oral bovine lactoferrin (bLF), through its antimicrobial, antioxidant and anti-inflammatory properties, will reduce the rate of mortality or major morbidity in very low birth weight (VLBW) preterm infants.

DETAILED DESCRIPTION:
Almost 3,000 very low birth weight (VLBW), <1500g preterm infants are born and treated in Canada annually. About 1,200 either die or survive with severe brain or lung injury, retinopathy, late-onset sepsis or necrotizing enterocolitis (NEC), each of which is associated with substantial risk of childhood disability.

Lactoferrin is an antimicrobial, antioxidant, anti-inflammatory iron-carrying, bifidogenic glycoprotein found in all vertebrates and in mammalian milk, leukocytes and exocrine secretions. However, most VLBW infants receive insufficient human lactoferrin (hLF) from human breast milk in the first months of life, resulting in suboptimal protection. Because hLF is expensive, bovine lactoferrin (bLF) has been considered as an alternate supplement to improve this suboptimal protection.

LIFT is one of several ongoing trials using higher doses of bovine bLF in the VLBW population (120-200 mg/kg/d). If LIFT confirms a 19% reduction in the relative risk of its primary outcome, bLF will have a major impact, translating into thousands more intact survivors without major morbidity in Australia, New Zealand, Canada, Europe and worldwide each year. As >90% of very preterm survivors at hospital discharge reach adulthood, this represents more than 19,000 life-years gained in Canada alone each year, one of the largest gains in intact survival in any specialty since neonatal surfactant and antenatal steroids

ELIGIBILITY:
An infant will be able to participate once a parent or guardian has provided a written informed consent and the infants must meet all of the following inclusion criteria:

* <1500 g at birth
* 2-7 days old and not moribund
* infant is considered to be stable by the clinical care team
* has initiated feeds

Any infant meeting any of the following exclusion criteria will be excluded from participation in this study

* severe congenital anomalies which are likely to cause death or known to contribute to an adverse neurodevelopmental outcome
* major congenital gastrointestinal anomalies which will prevent an early approach to feeding
* parents unable to provide informed consent

Ages: 2 Days to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 453 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
Hospital mortality or major morbidity | Randomization to 36 weeks corrected gestation or to transfer/discharge if earlier.
  Hospital mortality or major morbidity at 36 weeks corrected gestation defined as:
  * Brain injury on ultrasound
  * Necrotizing enterocolitis (Bell stage II or higher )
  * Late onset sepsis (≥ 72 hours of life, culture proven), or
  Retinopathy of prematurity treated according to local guidelines before discharge from hospital.

SECONDARY OUTCOMES:
Incidence of all-cause in-hospital mortality | Randomization to 36 weeks corrected gestation or to transfer/discharge if earlier
Incidence of each of the 5 components of the composite primary endpoint | Randomization to 36 weeks corrected gestation or to transfer/discharge if earlier
Incidence of chronic lung disease at 36 weeks CG | Randomization to 36 weeks corrected gestation or to transfer/discharge if earlier
Time to first day of full enteral feeds (≥120ml/kg/day for 3 consecutive days) | Randomization to 36 weeks corrected gestation or to transfer/discharge if earlier
Number of blood transfusions | Randomization to 36 weeks corrected gestation or to transfer/discharge if earlier
Length of hospital stay | Randomization to 36 weeks corrected gestation or to transfer/discharge if earlier
Weight and head circumference at 36 weeks corrected gestation | Randomization to 36 weeks corrected gestation or to transfer/discharge if earlier
Incidence of death by 24 months corrected age or the presence of neurodevelopmental outcomes at 24 months corrected age | Randomization to 36 weeks corrected gestation
  Incidence of death by 24 months corrected age or the presence of major neurodevelopmental outcomes at 24 months corrected age, as defined: (i) visual (cannot fixate/ legally blind, or corrected acuity <6/60 in both eyes), or hearing impairment (requiring a hearing aid or cochlear implants); (ii) cerebral palsy with an inability to walk unassisted; (iii) major developmental delay involving cognition or speech (composite score < 85 for cognition or language on assessment)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Asztalos, MD,MSc,FRCPC, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (9):
- Canada (9):
  - Foothills Medical Centre, Calgary, Alberta
  - Children's and Women's Health Centre BC, Vancouver, British Columbia
  - Health Sciences Centre Winnipeg, Winnipeg, Manitoba
  - Saint Boniface Hospital, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital, Hamilton, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schmidt B, Asztalos EV, Roberts RS, Robertson CM, Sauve RS, Whitfield MF; Trial of Indomethacin Prophylaxis in Preterms (TIPP) Investigators. Impact of bronchopulmonary dysplasia, brain injury, and severe retinopathy on the outcome of extremely low-birth-weight infants at 18 months: results from the trial of indomethacin prophylaxis in preterms. JAMA. 2003 Mar 5;289(9):1124-9. doi: 10.1001/jama.289.9.1124. PMID 12622582
- [Background] Bassler D, Stoll BJ, Schmidt B, Asztalos EV, Roberts RS, Robertson CM, Sauve RS; Trial of Indomethacin Prophylaxis in Preterms Investigators. Using a count of neonatal morbidities to predict poor outcome in extremely low birth weight infants: added role of neonatal infection. Pediatrics. 2009 Jan;123(1):313-8. doi: 10.1542/peds.2008-0377. PMID 19117897
- [Background] Schulzke SM, Deshpande GC, Patole SK. Neurodevelopmental outcomes of very low-birth-weight infants with necrotizing enterocolitis: a systematic review of observational studies. Arch Pediatr Adolesc Med. 2007 Jun;161(6):583-90. doi: 10.1001/archpedi.161.6.583. PMID 17548764
- [Background] Lonnerdal B. Nutritional roles of lactoferrin. Curr Opin Clin Nutr Metab Care. 2009 May;12(3):293-7. doi: 10.1097/MCO.0b013e328328d13e. PMID 19318940
- [Background] Albera E, Kankofer M. Antioxidants in colostrum and milk of sows and cows. Reprod Domest Anim. 2009 Aug;44(4):606-11. doi: 10.1111/j.1439-0531.2007.01027.x. PMID 19642220
- [Background] Embleton NE, Pang N, Cooke RJ. Postnatal malnutrition and growth retardation: an inevitable consequence of current recommendations in preterm infants? Pediatrics. 2001 Feb;107(2):270-3. doi: 10.1542/peds.107.2.270. PMID 11158457
- [Derived] Asztalos EV, Barrington K, Lodha A, Tarnow-Mordi W, Martin A. Lactoferrin infant feeding trial_Canada (LIFT_Canada): protocol for a randomized trial of adding lactoferrin to feeds of very-low-birth-weight preterm infants. BMC Pediatr. 2020 Jan 29;20(1):40. doi: 10.1186/s12887-020-1938-0. PMID 31996186
- See also: Canadian Neonatal Network. Accessed September 30, 2016. — http://www.canadianneonatalnetwork.org